CLINICAL TRIAL: NCT06769503
Title: Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University
Brief Title: Effect of Aromatherapy on Anxiety in Relatives of Emergency Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, principal investigator, Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Okutan2
Record Dates: First submitted 2025-01-05; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Emergency Service, Hospital; Aromatherapy; Anxiety
Keywords: emergency department; aromatherapy; anxiety
MeSH Terms: conditions — Emergencies; Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled experimental study in a pre-test-post-test control group experimental model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention Group After the patient is registered in the emergency department, the participant introduction form and state-trait anxiety scales will be applied as a pre-test to the relatives of the patient who agree to participate in the study. The participants will be made to smell lavender oil dropped on gauze by the researchers for an average of 3-5 minutes. The state and trait anxiety scales will be applied as a post-test approximately 15 minutes after the intervention.
  Interventions: Other: aromatherapy
- Control Group (No Intervention): Control Group After the patient is registered in the emergency department, the participant introduction form and state-trait anxiety scales will be applied as a pre-test to the relatives of the patient who agree to participate in the study. No intervention will be made to the control group participants. After a certain waiting period (average of 15 minutes), the state and trait anxiety scales will be applied as a post-test.

INTERVENTIONS:
Other: aromatherapy — Lavender oil dropped on gauze will be smelled for approximately 3-5 minutes.
  Arms: Intervention Group

SUMMARY:
This study aims to determine the effect of aromatherapy (lavender oil) application on the anxiety level of relatives of patients admitted to the emergency department.

The hypotheses of the study are as follows:

H1: Aromatherapy (lavender oil) application has an effect on the anxiety level of relatives of patients presenting to the emergency department.

H0: Aromatherapy (lavender oil) application has no effect on the anxiety level of relatives of patients presenting to the emergency department.

DETAILED DESCRIPTION:
In the experimental group; After the patient is registered in the emergency department, the participant introduction form and state-trait anxiety scales will be applied as a pre-test to the relatives of the patients who agree to participate in the study. The participants will be made to smell lavender oil dropped on gauze by the researchers for an average of 3-5 minutes. After the intervention, the state and trait anxiety scales will be applied as a post-test approximately 15 minutes later.

In the control group; After the patient is registered in the emergency department, the participant introduction form and state-trait anxiety scales will be applied as a pre-test to the relatives of the patients who agree to participate in the study. No intervention will be made to the participants in the control group. After a certain waiting period (after an average of 15 minutes), the state and trait anxiety scales will be applied as a post-test.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18 years of age or older
2. Not having a problem with smell
3. Accompanying the patient
4. Not having a psychiatric problem

Exclusion Criteria:

1. Refusing to participate in the study or wanting to leave
2. Having an upper respiratory tract infection
3. Known history of allergy (lavender oil)
4. Having a chronic respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
anxiety level | It will take approximately 30 minutes.
  The anxiety levels of patients will be measured using the "State and Trait Anxiety Scale".
  State and Trait Anxiety Scale; consists of two scales. Each scale has 20 questions. Scoring is between 1-4. Each scale score varies between 20-80 points. A high scale score indicates high anxiety. A low scale score indicates low anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin OKUTAN, Dr., Principal Investigator — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)